CLINICAL TRIAL: NCT00247988
Title: Phase II Study of Weekly Carboplatin and Taxotere in Platinum Sensitive Relapsed Ovarian or Tubal or Primary Peritoneal Cancers
Brief Title: Weekly Carboplatin and Taxotere in Platinum Sensitive Relapsed Ovarian or Tubal or Primary Peritoneal Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Regulatory issues(trial temporarily suspended December 28, 2005. Permanently suspended January 19, 2007. Institutional Reveiw Board informed April 18, 2007
Sponsor: University of Saskatchewan (Other)
Collaborators: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRP69761/6021
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Platinum Sensitive Relapsed Ovarian Cancer
Keywords: Ovarian; Relapsed
MeSH Terms: conditions — Recurrence

INTERVENTIONS:
Drug: Weekly Taxotere with weekly carboplatin

SUMMARY:
Weekly carboplatin and taxotere will be tolerable and effective as second line treatment of platinum-sensitive ( >6 month treatment free interval) relapsed ovarian cancer

Primary efficacy parameter will be response rate (CR and PR) according to RECIST criteria.

Secondary endpoints will be duration of response, progression free survival and overall survival. Toxicity will also be evaluated.

DETAILED DESCRIPTION:
Ovarian cancer is the sixth most common malignancy in women, with estimated 2500 cases diagnosed in 2001, and 1500 deaths. Despite maximal cytoreductive therapy, followed normally by a taxane and carboplatin (or cisplatin) chemotherapy, most patients will relapse, and require chemotherapy in a palliative setting. The goal of this second line therapy is to prolong survival and to improve quality of life. This disease has been characterized as chronic, as many patients may eventually go on to respond to additional lines of therapy.

Response to second line therapy has been correlated to length of time since the end of the first line treatment (treatment free interval, TFI). Patients relapsing or progressing while on therapy are defined as platinum-refractory. In North America the norm is to label patients with a TFI of 6 months or less as platinum-resistant. A TFI of greater than 6 months would make a patient platinum-sensitive.

These platinum-sensitive patients are generally treated with single agent carboplatin or carboplatin and taxol by 3-weekly administration. The ICON-4 trial published in June 2003 compared single agent platinum to combination of platinum-taxol. Patients could have received one or both of these agents in the adjuvant setting. At a median follow-up of 42 months the absolute difference in 2-year survival was 7% [P=0.0004} in favor of the combination arm. Thus combination platinum-taxol is the present standard of care in platinum-sensitive relapsed ovarian cancer. Use of taxol is limited by persistent neuropathy in 20%.

Presently there is growing evidence in support of giving chemotherapy at shorter intervals at low-doses. Hypothetically, this allows less advancement of cancer cells through the cell cycle. Moreover weekly taxanes are associated with an anti-angiogenic effect- more so with taxotere than taxol in cell-lines.

Several randomized trials in breast cancer have shown the improved efficacy of weekly taxol over 3-weekly taxol. The neoadjuvant study showed an increase in pCR [complete response on pathologic evaluation] of 10%with weekly taxol. The adjuvant study with 2-weekly chemotherapy showed a 7% improvement in time-to-progression over 3-weekly chemotherapy.

In ovarian cancer- a Phase II study of weekly carboplatin (AUC-2) with taxol (80mg/m2/week) given on day 1,8,15 of 28 day cycles has shown a response rate of 100% [80% CR, 20% PR] in 21 platinum-sensitive patients- with either measurable or evaluable disease. Median duration of response was 11.7 months (95% CI- 8.0-18.5 months). 46% reported Grade I neuropathy, 1 patient had febrile neutropenia, and 32% had Grade 3 neutropenia.

Weekly administration of taxotere with carboplatin has been studied in a Phase I study. Maximum tolerated dose was Taxotere 35mg/m2 with carboplatin AUC-2. At this dose no Grade 3 or 4 cytopenias were seen. Nor were there significant neuropathies.

Our study plans to evaluate Taxotere 35mg/m2 with Carboplatin at AUC-2 given weekly. 3 weekly treatments will constitute one cycle. We expect to see equivalent response rates and equivalent or higher duration of responses with better toxicity profile.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must demonstrate their willingness to participate in the study (reliable and compliant for repeated treatments) and comply with its procedures by signing a written informed consent.
2. Subjects must be 18 years of age or older.
3. Subjects must have received a platinum regimen, with or without paclitaxel or cyclophosphamide, and have maintained a disease-free status for at least 6 months following the completion of first line therapy.
4. Documented measurable or evaluable ovarian, tubal or primary peritoneal cancer by appropriate radiologic imaging (x-ray, or CT scan). Radiation therapy is allowed as long as not at the site of measurable disease. Recurrent disease based on elevated CA-125 alone is allowed, provided it meets the CA-125 progression definition.
5. Subjects must have adequate hepatic, renal and marrow function (AST/ALT< 3UNL, creatinine<2UNL, ANC>2, HGB>90)
6. Histologic diagnosis of ovarian, tubal or primary peritoneal cancer.
7. Performance status: ECOG Score greater than or equal to 2.
8. Subjects must have life expectancy of at least 6 months.
9. Women of childbearing potential must have a negative pregnancy test at time of enrollment and must be using an acceptable method of birth- control during the study.

Exclusion Criteria:

1. Female subjects who are pregnant, breast-feeding, or unwilling to use adequate contraception.
2. Any other active primary tumor under treatment, except basal cell carcinoma of the skin, or carcinoma in situ of the cervix;
3. Two or more prior chemotherapy regimens for ovarian cancer
4. Serious infection within one month of commencement of treatment.
5. Patients with known brain metastasis. However baseline CT of the head is not a must.
6. Patients with severe gastro-intestinal symptoms- e.g.- partial obstruction, bleeding or diarrhea.
7. Patients with Grade 2 or higher neuropathy [NCI Common toxicity criteria].

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38
Dates: Start 2003-10; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Response rate (CR and PR) according to RECIST criteria.

SECONDARY OUTCOMES:
Duration of response, progression free survival and overall survival. Toxicity will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: mohammed salim, MD, Study Chair — Saskatoon Cancer Center
Locations (1):
- Saskatoon Cancer Center, Saskatoon, Saskatchewan, Canada